CLINICAL TRIAL: NCT04721106
Title: A Prospective, Single-arm, Open-label, Non-interventional, Multi-centre, Post Marketing Surveillance (PMS) Study of Vizimpro®
Brief Title: Korea Post Marketing Surveillance (PMS) Study of Vizimpro
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A7471060; NCT04721106 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2021-01-13; First posted 2021-01-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Lung Neoplasms
Keywords: EGFR NSCLC
MeSH Terms: conditions — Lung Neoplasms | interventions — dacomitinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vizimpro treatment group: This group is included the patients that Vizimpro are prescribed and administrated according to local label in the routine clinical practice
  Interventions: Drug: Vizimpro

INTERVENTIONS:
Drug: Vizimpro — treatment group

SUMMARY:
Vizimpro will be approved for the treatment of EGFR NSLCL 1L in Korea. In accordance with the Standards for Re-examination of New Drug, it is required to conduct a PMS. Post marketing surveillance is required to determine any problems or questions associated with Vizimpro after marketing in Korea, with regard to the following clauses under conditions of general clinical practice. Therefore, through this study, effectiveness and safety of Vizimpro will be observed.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. Vizimpro® naïve patients to whom Vizimpro® can be prescribed as per the local labeling (the first-line treatment of adult patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) with epidermal growth factor receptor (EGFR) exon 19 deletion or exon 21 L858R substitution mutations
2. Evidence of a signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study

Exclusion criteria

Patients meeting any of the following criteria will not be included in the study:

1. Patients to whom Vizimpro® is contraindicated as per the local labeling. A. Hypersensitivity to the active substance or to any of the excipients of this product.

   B. This medicinal product contains lactose. Patients with rare hereditary conditions of galactose intolerance, total lactase deficiency, or glucose-galactose malabsorption should not take this medicinal product.
2. Any patients (or a legally acceptable representative) who does not agree that Pfizer and companies working with Pfizer use his/her information.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients to whom Vizimpro can be prescribed as per the local labeling (the first-line treatment of adult patients with locally advanced or metastatic NSCLC with epidermal growth factor receptor EGFR-activating mutations
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2021-03-07 (Actual); Primary Completion 2026-01-19 (Actual); Study Completion 2026-01-19 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events categorized according to physical organ and disease/symptom | From Day 1 of first administration dose up to the date of at least 28 calendar days following the last administration

SECONDARY OUTCOMES:
overall response rate | Day 1 until progression or drop out of study
  This study is observation, non-intervention study in routine clinical practice. Response rate according to RECIST criteria will be collected under routine clinical practice visit.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A7471060